CLINICAL TRIAL: NCT05448521
Title: Association of Postoperative Lactate Levels With Postoperative Atrial Fibrillation in Patients Undergoing Isolated Coronary Artery Bypass Graft Surgery
Brief Title: Postoperative Lactate and Atrial Fibrillation After CABG
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Başakşehir Çam & Sakura City Hospital (Other Government)
Responsible Party: Principal Investigator, Zeki Temiztürk, Principal Investigator, Başakşehir Çam & Sakura City Hospital
Other Study IDs: KAEK/2021.12.289
Record Dates: First submitted 2022-07-01; First posted 2022-07-07 (Actual); Last update posted 2022-10-10 (Actual); Status verified 2022-10

CONDITIONS: Coronary Artery Disease; Atrial Fibrillation
MeSH Terms: conditions — Coronary Artery Disease; Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Low lactate: Patients with a low lactate level defined by logistic regression analysis.
- High lactate: Patients with a high lactate level defined by logistic regression analysis.

SUMMARY:
Postoperative atrial fibrillation (POAF) is associated with increased mortality and morbidity in patients undergoing isolated coronary artery bypass grafting (CABG). It has been estimated that 5-40% of CABG patients experience POAF. Advanced age, P wave abnormalities, left atrial dilation, emergency surgery, low left ventricle ejection fraction, low glomerular filtration rate and chronic obstructive pulmonary disease have been reported in the etiology. Predicting which patients would experience POAF following CABG is important since it would allow physicians to apply more focused prophylactic measures. Lactate is the final product of anaerobic glycolysis. Serum lactate level are increased in case of inadequate oxygen delivery to tissues. The investigators aim to assess whether serum lactate levels measured early in the postoperative period could be used as a predictive marker of POAF in adults undergoing isolated CABG.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing isolated CABG
* Age >18 years

Exclusion Criteria:

* Age <18 years
* Pregnancy
* History of paroxysmal atrial fibrillation prior to surgery
* Undergoing concomitant procedures (e.g., CABG + valve surgery)
* Any preoperative cardiac rhythm other than normal sinus rhythm
* More than mild cardiac valve stenosis or insufficiency

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All consecutive adult patients undergoing isolated CABG during the study period in the Department of Cardiovascular Surgery at Basaksehir Cam Sakura City Hospital will be evaluated for possible enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2022-08-15 (Actual); Primary Completion 2023-08-15 (Estimated); Study Completion 2023-09-15 (Estimated)

PRIMARY OUTCOMES:
Postoperative atrial fibrillation | 30 days
  New-onset atrial fibrillation occurring in the immediate period after CABG

CONTACTS AND LOCATIONS:
Overall Officials: Ahmet Can Topcu, MD, Principal Investigator — Başakşehir Çam & Sakura City Hospital
Locations (1):
- Basaksehir Cam Sakura City Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Greenberg JW, Lancaster TS, Schuessler RB, Melby SJ. Postoperative atrial fibrillation following cardiac surgery: a persistent complication. Eur J Cardiothorac Surg. 2017 Oct 1;52(4):665-672. doi: 10.1093/ejcts/ezx039. PMID 28369234
- [Background] O'Connor E, Fraser JF. The interpretation of perioperative lactate abnormalities in patients undergoing cardiac surgery. Anaesth Intensive Care. 2012 Jul;40(4):598-603. doi: 10.1177/0310057X1204000404. PMID 22813486
- [Background] Dobrev D, Aguilar M, Heijman J, Guichard JB, Nattel S. Postoperative atrial fibrillation: mechanisms, manifestations and management. Nat Rev Cardiol. 2019 Jul;16(7):417-436. doi: 10.1038/s41569-019-0166-5. PMID 30792496